CLINICAL TRIAL: NCT04101825
Title: Open, Non-comparative Study to Evaluate the Performance and Safety of the Medical Device AURALYA® (Hyaluronic Acid-dermal Filler) in the Treatment of Nasolabial Wrinkles to Obtain Facial Rejuvenation
Brief Title: MD Auralia (HA Filler) in Treatment of Nasolabial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPIRA/0219/MD
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Nasolabial Fold, Hypoplastic

STUDY DESIGN:
Intervention Model Description: This trial is open label, multi-center, non-randomized single group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auralya (Experimental): Auralya® 25 (Cross-linked Hyaluronic Acid) Injection
  Interventions: Device: Auralya

INTERVENTIONS:
Device: Auralya — Hyaluronic Acid-Dermal Filler

SUMMARY:
Auralya® is a sterile, injectable, non-pyrogenic, re-absorbable medical product made of reticulated hyaluronic acid of non-animal origin, produced via bacterial fermentation.

To evaluate the overall safety of the medical device and performance of Auralya® dermal filler in terms of absolute change of WSRS score (Wrinkle Severity Rating Scale) assessed by Investigator at 8 and 12 weeks after the initiation of treatment, compared to Baseline Visit (day 0).

DETAILED DESCRIPTION:
Minimally invasive procedures (injectable dermal fillers) are among the techniques preferred by an increasing number of specialists in Aesthetics due to their clinical performance regarding volume restoration, and favourable safety profile.

During January - March 2018, it was performed a review of the scientific literature to find similar investigations to determine the minimal clinical significant difference between Baseline and a period of 30 days after the end the treatment.

In a similar dermal filler study, Takanobu Mashiko et al used a 5-grade WSRS and showed that, at 4 weeks after treatment, they achieved a 1.7 ± 0.5 (mean ± SD) improvement between those visits.

Considering the exploratory nature of this study and the fact that this investigation is first in-human, we choose to take a 0.5 WSRS decrease, at 90 days from the treatment start, as a minimal clinically significant difference. The standard deviation considered for the sample size calculation was set at 0.8 WSRS points.

By using a one-sided Wilcoxon Signed-rank test (matched pairs), a significance level of 0.05 and a power of 0.95 (probability of finding an effect when there is one), we calculated a total sample size of 31 subjects.

ELIGIBILITY:
Inclusion criteria:

1. Men or women with age > 35 and ≤ 65 years.
2. Subjects with nasolabial wrinkles, seeking tissue augmentation treatment and willing to receive HA Filler;
3. Subjects presenting a score of 2 (shallow wrinkles) or 3 (moderate, deep wrinkles) on the Wrinkles Severity Ranking Scale (WSRS);
4. Subjects who agree to discontinue all dermatological treatment and procedures during the study;
5. Subjects willing to provide signed informed consent to clinical investigation participation.
6. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Exclusion criteria:

1. Subjects who have bleeding disorder in the past or present.
2. Use of aspirin and antiplatelet agents a week prior to treatment
3. Prior or planned use of topical injection to the face (steroid, retinoid: applicable only to drugs, not applicable to cosmetics), within 4 weeks prior to screening or during this study (steroid ointment for therapeutic objectives is allowed for short -term use of ≤14 consecutive days.).
4. Use of immunosuppressive, chemotherapies, or systemic corticosteroids within 12 weeks from screening.
5. History of anaphylaxis or severe complicated allergy symptoms.
6. Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders or previous mental disorders that may significantly affect the study.
7. Hypersensitivity skin reaction to the investigational device based on intradermal test results at screening.
8. Evidence or history of autoimmune disease or compromised immune system.
9. Treatment with anticoagulants, thrombolytics, or platelet inhibitors within 1 week prior to study participation;
10. Prior permanent fillers or fat graft procedures around nasolabial folds.
11. Wrinkle correction procedures (e.g., botulinum toxin A injection, face lift, soft tissue augmentation, medium-depth peel, dermal photorejuvenation, etc.) within 6 months prior to study participation.
12. History of hypersensitivity to local anesthetic of amide type or HA.
13. History of keloid formation or hypertrophic scar on the face.
14. Evidence of active infection on the face.
15. Wound, scar, or skin disorder or infection around nasolabial folds that may affect the efficacy assessment.
16. Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study, *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
17. As with all dermal filler procedures, the product should not be used in vascular rich areas.
18. Subjects with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the study.
19. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and performance of Auralya | 12 weeks
  To evaluate the overall safety of the medical device and performance of Auralya® dermal filler in terms of absolute change of Wrinkle Severity Rating Scale assessed by Investigator at 8 and 12 weeks after the initiation of treatment, compared to Baseline Visit (day 0).

SECONDARY OUTCOMES:
Change of Wrinkle Severity Rating Scale | 12 weeks
  Absolute change of WSRS score assessed by the subject at 2, 4, 8 and 12 weeks compared to Baseline Visit (day 0).
General appearance after treatment | 12 weeks
  General appearance after treatment assessed by the subject at 2, 4, 8 and 12 weeks after the first treatment session compared to Baseline Visit (day 0) using the Global Aesthetic Improvement Scale (GAIS)
Subject satisfaction | 12 weeks
  Subject satisfaction assessed at 2, 4, 8 and 12 weeks, through Treatment Satisfaction Questionnaire completed by the subject providing their degree of satisfaction with the treatment on a three-point scale (very satisfied, satisfied, or not satisfied)
Global evaluation of product performance | 12 weeks
  Global evaluation of product performance by Investigator with photos taken at each visit. The photos will be compared in the final visit (week 12)
Product safety | 12 weeks
  Global evaluation of product safety by Investigator and by the patient using Patient Global Assessment of Safety questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Fratila, MD, Principal Investigator — SCM Dr. Rosu
Locations (1):
- SCM Dr. Rosu, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Fitzgerald R, Graivier MH, Kane M, Lorenc ZP, Vleggaar D, Werschler WP, Kenkel JM. Update on facial aging. Aesthet Surg J. 2010 Jul-Aug;30 Suppl:11S-24S. doi: 10.1177/1090820X10378696. PMID 20844296
- [Background] Sudha PN, Rose MH. Beneficial effects of hyaluronic acid. Adv Food Nutr Res. 2014;72:137-176. doi: 10.1016/B978-0-12-800269-8.00009-9. PMID 25081082
- [Background] Kim BW, Moon IJ, Yun WJ, Chung BY, Kim SD, Lee GY, Chang SE. A Randomized, Evaluator-Blinded, Split-Face Comparison Study of the Efficacy and Safety of a Novel Mannitol Containing Monophasic Hyaluronic Acid Dermal Filler for the Treatment of Moderate to Severe Nasolabial Folds. Ann Dermatol. 2016 Jun;28(3):297-303. doi: 10.5021/ad.2016.28.3.297. Epub 2016 May 25. PMID 27274627
- [Background] Kopera D, Palatin M, Bartsch R, Bartsch K, O'Rourke M, Holler S, Baumgartner RR, Prinz M. An open-label uncontrolled, multicenter study for the evaluation of the efficacy and safety of the dermal filler Princess VOLUME in the treatment of nasolabial folds. Biomed Res Int. 2015;2015:195328. doi: 10.1155/2015/195328. Epub 2015 Mar 3. PMID 25821787
- [Background] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448
- [Background] Dong J, Gantz M, Goldenberg G. Efficacy and safety of new dermal fillers. Cutis. 2016 Nov;98(5):309-313. PMID 28040813
- [Background] De Boulle K, Heydenrych I. Patient factors influencing dermal filler complications: prevention, assessment, and treatment. Clin Cosmet Investig Dermatol. 2015 Apr 15;8:205-14. doi: 10.2147/CCID.S80446. eCollection 2015. PMID 25926750
- [Background] Rivkin AZ. Volume correction in the aging hand: role of dermal fillers. Clin Cosmet Investig Dermatol. 2016 Aug 30;9:225-32. doi: 10.2147/CCID.S92853. eCollection 2016. PMID 27621659
- [Background] Kuhne U, Esmann J, von Heimburg D, Imhof M, Weissenberger P, Sattler G. Safety and performance of cohesive polydensified matrix hyaluronic acid fillers with lidocaine in the clinical setting - an open-label, multicenter study. Clin Cosmet Investig Dermatol. 2016 Oct 20;9:373-381. doi: 10.2147/CCID.S115256. eCollection 2016. PMID 27799807
- [Background] Lorenc ZP, Bank D, Kane M, Lin X, Smith S. Validation of a four-point photographic scale for the assessment of midface volume loss and/or contour deficiency. Plast Reconstr Surg. 2012 Dec;130(6):1330-1336. doi: 10.1097/PRS.0b013e31826d9fa6. PMID 23190816
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] McCall-Perez F, Stephens TJ, Herndon JH Jr. Efficacy and tolerability of a facial serum for fine lines, wrinkles, and photodamaged skin. J Clin Aesthet Dermatol. 2011 Jul;4(7):51-4. PMID 21779421
- [Background] Rzany B, Cartier H, Kestemont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC, Ma YM. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol Surg. 2012 Jul;38(7 Pt 2):1153-61. doi: 10.1111/j.1524-4725.2012.02470.x. PMID 22759252
- [Background] Van Dyke S, Hays GP, Caglia AE, Caglia M. Severe Acute Local Reactions to a Hyaluronic Acid-derived Dermal Filler. J Clin Aesthet Dermatol. 2010 May;3(5):32-5. PMID 20725567
- [Background] Funt D, Pavicic T. Dermal fillers in aesthetics: an overview of adverse events and treatment approaches. Plast Surg Nurs. 2015 Jan-Mar;35(1):13-32. doi: 10.1097/PSN.0000000000000087. PMID 25730536
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Yeom J, Bhang SH, Kim BS, Seo MS, Hwang EJ, Cho IH, Park JK, Hahn SK. Effect of cross-linking reagents for hyaluronic acid hydrogel dermal fillers on tissue augmentation and regeneration. Bioconjug Chem. 2010 Feb 17;21(2):240-7. doi: 10.1021/bc9002647. PMID 20078098
- [Background] Jiang LI, Stephens TJ, Goodman R. SWIRL, a clinically validated, objective, and quantitative method for facial wrinkle assessment. Skin Res Technol. 2013 Nov;19(4):492-8. doi: 10.1111/srt.12073. Epub 2013 Jun 10. PMID 23750828
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957